CLINICAL TRIAL: NCT03641924
Title: Cognition and Psychotherapy in PTSD: Mechanisms and Functional Outcomes
Brief Title: Cognition and Psychotherapy in PTSD
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D2699-R
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Posttraumatic Stress Disorder; Psychotherapy; Neuropsychology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PTSD: Veterans diagnosed with Diagnostic and Statistical Manual (DSM-V) PTSD
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is an evidence-based psychotherapy for PTSD.

SUMMARY:
Posttraumatic stress disorder (PTSD) is prevalent among combat Veterans and is a substantial public health burden. Several psychotherapies, including cognitive processing therapy (CPT) and prolonged exposure therapy, have been recommended as efficacious for the treatment of PTSD and are being disseminated nationally in the VA Healthcare System. Yet many individuals show limited benefit from such treatments. Accumulating evidence indicates that episodic memory deficits may be one factor limiting psychotherapy treatment efficacy in PTSD. The proposed study will determine whether verbal memory is a specific predictor of CPT outcomes in PTSD, including both symptom reductions and functional outcomes. The study will also determine the pathways by which memory functioning affects treatment outcomes by examining relationships between memory functioning, treatment engagement, recall of treatment content, and illness course. More specifically, analyses will examine whether memory for treatment content affects the relationship between memory functioning and treatment outcomes.

DETAILED DESCRIPTION:
Accumulating evidence indicates that memory dysfunction: 1) is prominent in PTSD; and 2) adversely affects psychotherapy outcomes. Identifying mechanisms underlying the relationship between memory dysfunction and poor treatment outcomes is crucial to provide empirical guidance regarding appropriate rehabilitation targets to reduce the impact of cognitive dysfunction on therapy outcomes.

In this study, the investigators aim to examine the specific effects of verbal memory on both PTSD symptoms and functional outcomes during CPT (Aim 1); identify the pathways by which cognitive dysfunction affects psychotherapy treatment response, with a focus on memory for treatment content and treatment adherence (Aim 2).

To achieve these aims, the investigators will enroll 105 Veterans with PTSD, who will complete a standard course of cognitive processing therapy (CPT) and complete longitudinal assessments of PTSD symptoms, functional status, treatment adherence, and memory for treatment content. This study does not randomize participants to treatment since all participants will be initiating CPT.

Recruitment. Participants will primarily be drawn from clinical referrals for PTSD therapy at the Corporal Michael J. Crescenz VA Medical Center (CMC VAMC) or its Community Based Outpatient Clinics (CBOCs).

Procedures. Participants will provide written informed consent and undergo intake screening. Major assessments will be conducted with participants at study entry (baseline), after session 6, and after session 12 (critical endpoint assessment) of CPT.

Baseline Visit (180-240 mins). Baseline procedures (before starting CPT) include diagnostic interviews, questionnaires assessing mood and functioning, a neurocognitive assessment, and additional memory measures. Participants will complete structured interview assessments for psychiatric conditions including PTSD, stressful life events, sociodemographics and medical history, and traumatic brain injury. Self-report assessments of mood, functional status (e.g., social adjustment), combat exposure, and behavioral functioning will also be administered. The neurocognitive assessment will include conventional neuropsychological tests and tests drawn from the Penn Computerized Neurocognitive Battery to assess multiple cognitive domains including memory, attention, speed of information processing, executive functioning, social cognition, and an IQ estimate. Additional experimental measures of memory processes from cognitive science will also be administered.

Psychotherapy. After the baseline visit, participants will begin a standard course of CPT (12 sessions) following standardized protocols (Resick et al, 2008) with the investigators' study therapists, who will all have extensive, formalized training in CPT and be supervised by an expert in CPT. Therapists will be blinded to scores on cognitive measures. After the initial CPT session, participants will complete questionnaires of treatment expectancy and self-efficacy (10 mins). At every following CPT visit, patients will complete brief questionnaires of adherence and application of treatment, depression symptoms, and suicide risk.

Mid-Treatment Assessments (20-30 mins). At CPT sessions 4, 6, 8, and 12 (end), participants will complete measures of memory for treatment content, treatment expectancy, and brief re-assessments of PTSD, mood, and functioning.

End of Treatment Assessment (120-180 mins). At the end of treatment, a final visit will consist of questionnaires and interviews to assess symptoms of PTSD, mood, functioning, cognitive functioning and memory for treatment content.

Although not a clinical trial, the investigators will examine individual change in symptoms at treatment end. Participants who drop out and are not able to be re-engaged will be contacted by study staff and asked to participate in a final assessment. After this visit is complete (or if the participant refuses), Veterans will be offered additional treatment at CMC VAMC as appropriate, with a warm handoff from study staff to the clinical team. Treatment non-responders, defined as participants displaying less than a 10-point reduction in CAPS Scores at follow-up, will also be referred for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 criteria for PTSD via the Clinician Administered PTSD Scale (CAPS-5)
* Willing to initiate CPT

Exclusion Criteria:

* Substance use disorder (moderate or above) not in remission for >1 mo
* Severe psychiatric illness (e.g., psychosis)
* Significant current suicidal or homicidal intent, including a specific plan
* Dementia, neurological disorder, or severe traumatic brain injury (TBI; i.e., loss of consciousness > 24h)
* Inability to speak or read English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Scott, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets will be shared upon written request. The PI and his team will create de-identified, study-specific dataset, replacing identifying information with study-specific codes. Investigators requesting access to a dataset will be asked to sign a Letter of Agreement or Data Use Agreement that will need to be approved by the local VA Information Security Officers and Privacy Officer. The investigators will follow specific VA Office of Research & Development Guidance.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Datasets meeting VA standards for disclosure to the public will be made available within one year of publication of primary results.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants either did not meet criteria for PTSD after a structured assessment (n=19), met criteria for a comorbid disorder that was exclusionary (n=4), or were lost to follow-up before completing baseline assessments.
Groups:
- Posttraumatic Stress Disorder (PTSD): Veterans diagnosed with DSM-V PTSD
  Cognitive Processing Therapy: Cognitive Processing Therapy is an evidence-based psychotherapy for PTSD.
Period: Overall Study
Arm/Group | Posttraumatic Stress Disorder (PTSD)
Started | 110 (Enrolled)
Received Intervention | 94
Completed | 58
Not Completed | 52
Not completed — Withdrawal by Subject | 26
Not completed — Lost to Follow-up | 16
Not completed — Protocol Violation | 10

BASELINE CHARACTERISTICS:
Groups:
- Veterans With PTSD: Veterans with DSM-5 PTSD as assessed with the Clinician Administered PTSD Scale
Arm/Group | Veterans With PTSD
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 40
  White | 45
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 94
Mild Traumatic Brain Injury (TBI) [Count of Participants; unit: Participants] | 49
Moderate TBI [Count of Participants; unit: Participants] | 7
PTSD Checklist (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — Range = 0-80; higher scores equal greater PTSD symptoms.
  units on a scale | 45 (11)

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Checklist (PCL-5)
Description: PTSD Symptoms. The range of the scale is from 0 (no symptoms) to 80 (maximal symptoms). Higher scores corresponds to more symptoms.
Time Frame: Change from baseline to 12 weeks
Population: Based on baseline memory scores
Measure: Mean (Standard Deviation); unit: change in units on a scale
Groups:
- Low Memory: Bottom tertile of memory performance
- Medium Memory: Middle tertile of memory performance
- High Memory: Top tertile of memory performance
Arm/Group | Low Memory | Medium Memory | High Memory
Number analyzed (Participants) | 31 | 32 | 31
change in units on a scale | 9.25 (20.37) | 11.94 (15.93) | 15.91 (15.10)

2. Primary Outcome: Social Adjustment Scale-Self Report (SAS-SR)
Description: Functional Status. Scored 1-5, with higher scores indicating worse functioning.
Time Frame: Change from baseline to 12 weeks
Population: Groups based on baseline memory scores
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Low Memory | Medium Memory | High Memory
Number analyzed (Participants) | 30 | 31 | 30
change in units on a scale | 0.14 (0.56) | 0.10 (0.41) | 0.38 (0.42)

3. Secondary Outcome: Veterans RAND 12 Item Health Survey Mental Component Summary (VR-12 MCS)
Description: Mental Health-Related Quality of Life. Scores range from 0-100; higher values indicate better mental health-related quality of life.
Time Frame: Change from baseline to 12 weeks
Population: Based on baseline memory scores
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Low Memory | Medium Memory | High Memory
Number analyzed (Participants) | 30 | 31 | 30
change in units on a scale | 1.26 (7.95) | 0.32 (9.05) | 0.39 (6.11)

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- PTSD: Veterans diagnosed with DSM-V PTSD
  Cognitive Processing Therapy: Cognitive Processing Therapy is an evidence-based psychotherapy for PTSD.
Arm/Group | PTSD
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT03641924/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03641924/ICF_001.pdf